CLINICAL TRIAL: NCT02581579
Title: Pilot Phase I Clinical Trial, Double-blind, Randomized, Placebo Controlled and Masked to Evaluate the Tolerability and Immunogenicity of Nyaditum Resae ® Probiotic Administered to Pediatric Population in Contact With Tuberculosis With or Without Latent Tuberculosis Infection
Brief Title: Study to Evaluate the Tolerability and Immunogenicity of Nyaditum Resae ® Probiotic Administered to Pediatric Population in Contact With Tuberculosis With or Without Latent Tuberculosis Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manresana de Micobacteriologia, SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NYADAPETRICS
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Tregs; Tolerance; Probiotic; Mycobacteria
MeSH Terms: conditions — Tuberculosis; Mycobacterium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nyaditum resae ® 10e5 of heat-killed Mycobacterium manresensis (Active Comparator): Nyaditum resae ® 10e5 of heat-killed Mycobacterium manresensis
  Interventions: Dietary Supplement: Nyaditum resae ® 10e5 of heat-killed Mycobacterium manresensis
- Placebo (Placebo Comparator): MANITOL CAPSULES
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nyaditum resae ® 10e5 of heat-killed Mycobacterium manresensis — Nyaditum resae ® 10e5 of heat-killed Mycobacterium manresensis, 1 capsule per day during 14
  Arms: Nyaditum resae ® 10e5 of heat-killed Mycobacterium manresensis
Other: Placebo — Placebo, 1 capsule per day during 14
  Arms: Placebo

SUMMARY:
This is a doble-blind, masked, compared with placebo clinical trial in pediatric population in contact with tuberculosis with or without tuberculosis infection. This trial aims to study the effect of the probiotic Nyaditum resae® at the level of specific Treg memory cells eight weeks after the first administration, and the global tolerability of the treatment.

Nyaditum resae® is a preparation in the form of capsules containing heat-killed environmental mycobacteria Mycobacterium manresensis. The overall objective of the study is the effect of Nyaditum resae® on immunity, which could reduce the risk of developing active tuberculosis.

DETAILED DESCRIPTION:
The incidence of tuberculosis is still a problem of the first magnitude. Every year 1.5 million people die; there are 10 million cases of illness and 100 million new infected. The growing problem of multi-resistance is to be added, remaining so prevalent: 700,000 patients, a figure that increases annually with 100,000 people. Prevention of tuberculosis is currently very difficult because it is a disease caused by a bacillus (Mycobacterium tuberculosis) that is transmitted by air: No risk factor for becoming infected has been identified and there is still no prophylactic vaccine that prevents from infection. One of the most characteristic aspects of tuberculosis is that the majority (90-95 %) of people without immunity alterations do not develop the disease after being infected. As for people who do develop the disease, it is still not known why they develop it.

A group of researchers from the Institut Germans Trias i Pujol recently discovered a mechanism that explains this trend. In short, what happens is that certain people create a too strong inflammatory response against tuberculosis bacillus, which ends up creating massive destruction of the tissue that is around the bacillus and brings the characteristic lesion of tuberculosis: tuberculous cavity.

This group of researchers was devising ways to "reeducate" the immune system against the bacillus not make it aggressive. And they did it using two instruments. The first one, an environmental mycobacteria, namely a bacillus of the family of mycobacteria tuberculosis, that usually lives in the water we drink, so that at a greater or lesser extent we already have it in our intestinal flora. The second, inducing a tolerant response, like we do when we eat food. To induce a tolerant response, low and repeated doses of the product make the immune system of the digestive duct "used to" their presence. Thus, when it becomes to find the product, the immune system reacts in a very light and balanced manner, avoiding excessive inflammatory responses. The clearest example is the fact that our immune system "is used" to feed proteins and generates no rejection answers found in the intestinal mucosa.

Hence comes the probiotic Nyaditum resae®, a preparation in the form of capsules, containing a heat-killed Mycobacterium manresensis and thus can generate a cross-immunity with the tuberculosis bacillus. By giving low and repeated dose to generate a tolerant response, which happens when there is an infection by Mycobacterium tuberculosis, so that a balanced immune response is triggered able to reduce the risk of developing active tuberculosis.

Tolerability of Nyaditum resae® has been studied in adults. Next step is to asses its behavior in pediatric population, since is a particularly vulnerable population in countries where there is a high incidence of this disease.

ELIGIBILITY:
Inclusion Criteria:

Child from a study of contact with tuberculosis. Obtaining informed consent from parents / mothers or guardians and, over 12 years, obtaining the consent of the child.

Child between 2 and 17 years (inclusive) on the day of obtaining informed consent.

Willingness to fulfill the requirements of the protocol.

Exclusion Criteria:

Active tuberculosis. Enrollment in another clinical trial or study with sanitary product involving invasive techniques.

Chronic administration of: methotrexate, azathioprine, cyclophosphamide, oral corticosteroids (≥500mg cumulative prednisone dose, or equivalent; inhaled or topical steroids are allowed) and other immunosuppressive therapies / immunomodulatory .

Administration of blood products or blood derivatives during the 6 months prior to randomization.

Vaccination in the month prior to randomization. Anticipation of receiving vaccines duration of the study.

Detection by the researcher lack of knowledge or willingness to participate and fulfill all the requirements of the protocol.

Any other finding that the investigator's opinion, could jeopardize the performance of the protocol or significantly influence the results or interpretation of the effects of probiotic.

Known immunodeficiencies. Pregnancy or breastfeeding. Hypersensitivity to mannitol

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-12-09 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Specific Treg memory cells at week 1 | From Baseline to Week 8
Proportion of patients presenting adverse events related to study treatment. | From Baseline to Week 8

SECONDARY OUTCOMES:
Proportion of participants presenting gastrointestinal adverse events related to study treatment. | Baseline to week 8
Proportion of participants presenting systemic adverse events related to study treatment. | Baseline to week 8

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Germans Trias I Pujol Hospital, Badalona, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Valle Hebron Hospital, Barcelona

REFERENCES:
- [Derived] Tukvadze N, Cardona P, Vashakidze S, Shubladze N, Avaliani Z, Vilaplana C, Cardona PJ. Development of the food supplement Nyaditum resae as a new tool to reduce the risk of tuberculosis development. Int J Mycobacteriol. 2016 Dec;5 Suppl 1(Suppl 1):S101-S102. doi: 10.1016/j.ijmyco.2016.09.073. Epub 2016 Nov 14. PMID 28043488